Date: 20/11/2020

Hypnotic intervention for women with chronic pelvic pain: a pilot randomized control trial.

NCT number: Not Available.

Authors:

Tiffany Brooks BPsych (Hons.) MPsych (Health) MAPS (Orchid ID: 0000-0003-0277-4563)1,2

Dr Rebecca Sharp BN, BHSc (Hons), Ph.D (Orchid ID: 0000-0003-3334-2990)1

Dr Susan Evans (Orchid ID: 0000-0003-0347-604X) FRANZCOG FFPMANZCA3

Sonia Scharfbillig BSc, BPhty (Hons), M Musc Sports Phsyio. (No orchid ID)4

Dr John Baranoff B.Sc.(Hons.), MClinPsych, Ph.D (Orchid ID: 0000-0003-2339-1895) 3,5

Professor Adrian Esterman PhD MSc BSc (hons) FACE DLSHTM (Orchid ID 0000-000107324-9171) 1

1. The University of South Australia, 2. Aware Women's Health in Adelaide, South Australia 3. University of Adelaide. 4. Pelvic Floor Health 5. Centre for Treatment of Anxiety and Depression.

Correspondence to be sent to:

Miss Tiffany Brooks

257 Melbourne Street, NORTH ADELAIDE SA 5006 Email: brota010@mymail.unisa.edu.au

## **Human Research Ethics Committee**



University of South Australia

**Clinical and Health Sciences** 

Consent Form

This project has been approved by the University of South Australia's Human Research Ethics Committee. If you have any ethical concerns about the project or questions about your rights as a participant please contact the Executive Officer of this Committee, Tel: +618 8302 6330; Email: <a href="mailto:humanethics@unisa.edu.au">humanethics@unisa.edu.au</a>.

| SECTION 1: CONTACT AND PROJECT DETAILS | |
|---|---|
| Researcher's Full Name | Tiffany Brooks |
| Contact Details | Brota010@mymail.unisa.edu.au |
| Supervisor's Name (students only) | Professor Adrian Esterman |
| Contact Details | Adrian.esterman@unisa.edu.au |
| Project Number | 202935 |
| Project Title | Hypnosis for women with Chronic Pelvic Pain: A pilot study |

## **SECTION 2: PARTICIPANT CERTIFICATION**

In signing this form, I confirm that:

- I have read the Participant Information Sheet, and the nature and the purpose of the research project has been explained to me. I understand and agree to take part.
- I understand that participation is voluntary and I can withdraw my responses at any time without reason up until one week after the study has concluded.
- I understand the nature of my involvement in the project.
- I understand that I may not directly benefit from taking part in the project.
- I understand that I can withdraw from the project at any stage and that this will not affect my status now or in the future.
- I confirm that I am over 18 years of age.
- I understand that while information gained during the project may be published, I will not be identified and my personal results will remain confidential, unless required by law.
- I understand the confidentiality limits when submitting responses online.

| Participant's Signature | Printed Name | Date |
|-------------------------------------|--------------|------|
| SECTION 3: RESEARCHER CERTIFICATION | | |

| SECTION 3: RESEARCHER CERTIFICATION | | |
|---|---|---|
| I have explained the study to the participant and consider that he/she understand what is involved. | | |
| Researcher Signature | Printed Name | Date |